CLINICAL TRIAL: NCT04848402
Title: A Study to Investigate the Safety and Tolerability of a Wearable On-body Delivery System, and Exploratory Assessment of Participant Response With an Autoinjector, Following Subcutaneous Injections of Placebo in Healthy Participants
Brief Title: A Device Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17770; H7K-MC-O005 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-Body Delivery System (OBDS)/Multiple Bolus Injector (Experimental): On-Body Delivery System (OBDS)/Multiple bolus injector used to administer placebo subcutaneously (SC).
  Interventions: Device: On-Body Delivery System (OBDS)/Multiple Bolus Injector; Drug: Placebo
- Single Auto Injector (Experimental): Single auto injector used to administer placebo SC.
  Interventions: Device: Single Auto Injector; Drug: Placebo

INTERVENTIONS:
Device: On-Body Delivery System (OBDS)/Multiple Bolus Injector — Used to administer placebo SC.
  Arms: On-Body Delivery System (OBDS)/Multiple Bolus Injector
Device: Single Auto Injector — Used to administer placebo SC.
  Arms: Single Auto Injector
Drug: Placebo — Administered SC.

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of two different devices that may be used to inject medication just under the skin. Participants will receive placebo; no active drug will be given. The study will last up to five weeks for each participant, including a one-week overnight stay in the study center.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or female participants as determined by medical history, laboratory tests, physical examination, 12-lead ECGs, and vital signs.
* Body mass index (BMI) within the range of 18 to 32 kilograms per meter squared (kg/m²)
* Female participants must not be pregnant, and must test negative for pregnancy
* Agree to video recording during each administration event using the autoinjector or bolus injector

Exclusion Criteria:

* Have known allergies to any components of the placebo or related compounds, or history of significant atopy, or known allergies or irritation to adhesives (e.g. skin adhesives, band aid)
* Have an abnormal blood pressure as determined by the investigator
* Have a history or presence of a bleeding disorder
* Have a history of any types of neuropathy, radiculopathy, or fibromyalgia that would affect perception in abdominal wall
* Have self-perceived dullness or loss-of-sensation on either side of the body or the abdomen
* Have any condition that could affect pain perception from an injection
* Have tattoos or scars over the abdomen, or other factors (eg, rash, excessive folds of skin) that, in the investigator's opinion, would interfere with injection-site assessments
* Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the trial
* Are currently using or intend to use painkillers, aspirin, or other nonsteroidal Anti-inflammatory drugs, anticoagulant or antiaggregant drugs, over-the-counter or prescription medication for pain or inflammation
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 2 months or 5 half-lives (whichever is longer) should have passed
* Are unwilling to stop alcohol consumption
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Are unwilling to abide by the tobacco restrictions
* Poor peripheral venous access
* Have a pacemaker and/or similar devices/other implantables

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Device | Baseline through day 7
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LABCORP, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No